CLINICAL TRIAL: NCT06665321
Title: Internet-based Affect Focused Psychodynamic Therapy for Neuroticism: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LINNEA
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Trait Neuroticism
Keywords: Trait neuroticism; Internet-delivered psychodynamic therapy; Internet Intervention

STUDY DESIGN:
Intervention Model Description: After recruitment finished, participants will be randomized to either IPDT treatment or wait-list control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based psychodynamic therapy (Experimental): The treatment consist of a 9 week long IPDT intervention based on Affect Phobia Therapy with weekly therapist support.
  Interventions: Behavioral: Internet-based psychodynamic therapy (IPDT)
- Wait-list control condition (No Intervention): Wait-list control condition, participants have the option to contact the treatment team in case of worsened symptoms.

INTERVENTIONS:
Behavioral: Internet-based psychodynamic therapy (IPDT) — The intervention is 9 week long with weekly modules that the participants work with while receiving weekly support from an assigned therapist.
  Arms: Internet-based psychodynamic therapy

SUMMARY:
The purpose of the study is to investigate if internet delivered affect-focused psychodynamic therapy (IPDT) leads to lowered levels of trait neuroticism compared to a wait-list control condition. The target group is adults (18+) who experience mild to moderate symptoms of anxiety and/or depression. The IPDT treatment consists of 8 modules that the participants will work with for 9 weeks, with therapist support. Participants will be recruited in Sweden with nationwide recruitment.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with the aim to investigate if IPDT leads to lowered levels of trait neuroticism. Participants will either be randomized to the treatment which is based on Affect Phobia Therapy or to a wait-list control. Participants will have weekly contact with a therapist who will provide feedback and support.

Primary outcome measure is trait neuroticism (measured on the 24-Item Neuroticism scale of the IPIP-NEO-120). Secondary outcome measures will include measures of anxiety, depression, quality of life, emotion regulation, and defense mechanism adaptiveness. Emotion regulation and short measure of anxiety and depressive symptoms will be collected weekly throughout the treatment period. Pre-treatment measurement, post-treatment measurement, weekly measure, and one-year follow up is planned to be collected through an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Score 5 points or more on either the PHQ-9 or GAD-7
* 18 years or older
* Ability to speak, read and write in Swedish
* Have access to the internet and a smartphone, computer or other device

Exclusion Criteria:

* Severe psychiatric or somatic illness that makes participation difficult or impossible
* Ongoing addiction
* Acute suicidality
* Other ongoing psychological treatment
* Recent (within the latest month) changes in the dose of psychotropic medication or planned change of dose during the treatment weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Neuroticism scale of the Maples et al (2014) IPIP NEO PI 120 Item representation | Change between baseline, end of treatment after nine weeks and follow-up at 12 months after treatment termination.
  Measure of trait neuroticism. Consists of 24 items. Each item is scored from 0-4 with a total range of 0-96. A higher score reflects a higher level of trait neuroticism.

SECONDARY OUTCOMES:
Eysenck Personality Questionnaire Revised - Shortform (EPQR-S) | Change between baseline, end of treatment after nine weeks and follow-up at 12 months after treatment termination.
  12-item measure of trait neuroticism. Each item is score yes or no. Range 0-12 with a higher score indicating higher levels of neuroticism.
Patient Health Questionnaire-9 | Change between baseline, end of treatment after nine weeks and follow-up at 12 months after treatment termination.
  Measure depressive symptoms. Consist of nine items, scored from 0-3. A higher score indicates more depressive symptoms.
Generalized Anxiety Disorder-7 | Change between baseline, end of treatment after nine weeks and follow-up at 12 months after treatment termination.
  Measures symptoms of anxiety. 7 items scored from 0-3, with a higher score indicating more anxiety symptoms.
Brunnsviken Brief Quality of life scale | Change between baseline, end of treatment after nine weeks and follow-up at 12 months after treatment termination.
  Measures quality of life. 12 items scored from 0-4. A higher score indicates higher quality of life.
Difficulties in Emotion Regulation Scale-16 | Change between baseline, end of treatment after nine weeks and follow-up at 12 months after treatment termination. Will be measured on a weekly basis during the 9 weeks of the intervention period.
  Measure of emotion regulation. Consists of 16 items scored from 1-5. A higher score indicates less adaptive emotion regulation.
Defense Mechanism Rating Scale - Self Report 30 | Change between baseline, end of treatment after nine weeks and follow-up at 12 months after treatment termination.
  Measures adaptiveness of defense mechanisms. Consists of 30 items scored from 0-4. A higher overall defense score (ODF) indicates more more adaptive defense mechanisms.
Patient Health Questionnaire - 4 | Change between baseline, end of treatment after nine weeks. Will be measured on a weekly basis during the intervention.
  Brief measurer of depressive and anxiety symptoms. Consists of 4 items, scored from 0-3. A higher score indicates more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping, Östergörland, Sweden

IPD SHARING:
Plan to Share IPD: Undecided